CLINICAL TRIAL: NCT04178590
Title: Effects of Application Injectable Platelet-Rich Fibrin (i-PRF) as Adjunct Therapy in the Initial Treatment of Periodontitis
Brief Title: Effect of Injectable Platelet-Rich Fibrin (i-PRF) in Initial Treatment of Chronic Periodontitis
Acronym: EIPRFITCP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Natasa Nikolic Jakoba, Associate professor, DDS, MSc, PhD, University of Belgrade
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UBelgrade 783/2
Record Dates: First submitted 2019-11-21; First posted 2019-11-26 (Actual); Results first posted 2020-06-11 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Periodontitis
Keywords: periodontitis; therapy; Platelet; Rich; Fibrin; Nonsurgical
MeSH Terms: conditions — Periodontitis | interventions — proliferation regulatory factors, human urine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: split mouth design
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SRP + Injectable Platelet-Rich Fibrin (Experimental): Scaling and root planing in conjunction with Injectable Platelet-Rich Fibrin
  Interventions: Drug: SRP + Injectable Platelet-Rich Fibrin
- SRP + placebo (Placebo Comparator): Scaling and root planing in conjunction with saline
  Interventions: Drug: SRP + placebo

INTERVENTIONS:
Drug: SRP + Injectable Platelet-Rich Fibrin — Injectable Platelet-Rich Fibrin application as adjunct to scaling and root planing
  Other Names: SRP + i-PRF
  Arms: SRP + Injectable Platelet-Rich Fibrin
Drug: SRP + placebo — Saline application during scaling and root planing
  Other Names: SRP + saline
  Arms: SRP + placebo

SUMMARY:
Current treatments of periodontitis have limited efficacy since they fail to suppress microorganisms satisfactorily over time. The aim of present study was to investigate whether there are differences between initial treatment of chronic periodontitis (SRP) and SRP in conjunction with injectable platelet-rich fibrin (i-PRF) application.

DETAILED DESCRIPTION:
Current treatments of periodontitis have limited efficacy since they fail to suppress microorganisms satisfactorily over time. The aim of present study was to investigate whether there are differences between initial treatment of chronic periodontitis (SRP) and SRP in conjunction with injectable platelet-rich fibrin (i-PRF) application.

Thirty patients with chronic periodontitis who had at least two sites with perriodontal pocket depth (PPD) ≥ 4 mm on contralateral side will be involved in the study. Using a split-mouth design, patients will be treated with SRP + I-PRF -(test group) or SRP only-(control group). Gingival crevicular fluid (GCF) and subgingival plaque will be collected with paper points (DentsplyMaillefer, Tulsa, Oklahoma, USA) at baseline and 1, 3 and 6 months after the treatment. The presence and concentrations of Aggregatibacter actinomycetemcomitans (Aa), Porphyromonas gingivalis (Pg), Prevotella intermedia (Pi) and Tannerella forsythia(Tf) will be analyzed by real-time polymerase chain reaction (qPCR). Periodontal parameters, including bleeding on probing (BOP), probing pocket depth (PPD) and the clinical attachment level (CAL), will be recorded on both sides, as well as concentration of TNF-alpha (tumor necrosis factor alpha), ALP(alkaline phosphatase) and MMP-8 (matrix-metalloproteinase-8).

ELIGIBILITY:
Inclusion Criteria:

* A minimum of 6 teeth per quadrant;

  * A minimum of 2 teeth in each quadrant with a probing depth (PD) ≥5 mm;
  * Bleeding on probing (BOP) had to be at ≥40% tooth sites;
  * No involvement of furcation;
  * Good general health.

Exclusion Criteria:

* Periodontal therapy within last 12 months;

  * Having surgical therapy;
  * Use of antibiotics over the last 6 months;
  * Ongoing drug therapy that might have an impact on the clinical signs and symptoms of periodontitis;
  * Pregnancy or nursing;
  * Current and former smokers.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mila Vuckovic, Dr., Principal Investigator — Assistant Lecturer
Locations (1):
- Department of Periodontology and Oral medicine, School of Dental Medicine, University of Belgrade, Belgrade, Serbia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: October 2019 Department of Periodontology and Oral Medicine School of Dental Medicine University of Belgrade
Pre-assignment Details: Periodontitis patients with systemic and/or other oral disease or ongoing drug therapy are excluded.
Units Other Than Participants: periodontal pockets
Groups:
- All Study Participants: Study participants randomly assigned to receive two different treatments in cross - over study design: Scaling and root planing in conjunction with Injectable Platelet-Rich Fibrin and Scaling and root planing in conjunction with saline
Period: Overall Study
Arm/Group | All Study Participants
Started ("split mouth" - both treatment modalities were conducted in all patients) | 32; 64 periodontal pockets
Completed | 30; 60 periodontal pockets
Not Completed | 2; 4 periodontal pockets
Not completed — Pregnancy | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: 32 participants
Units Other Than Participants: periodontal pocket
Groups:
- All Study Participants: Study participants randomly assigned to receive two different treatments in cross- over study design : scaling and root planing in conjunction with Injectable Platelet-Rich Fibrin and Scaling and root planing in conjunction with saline
Arm/Group | All Study Participants
Number analyzed (Participants) | 32
Number analyzed (periodontal pocket) | 64
Age, Categorical [Count of Participants; unit: Participants] — Population: unit was periodontal pocket - one side of the jaw (left or right), not whole patient
  Participants
    <=18 years | 0
    Between 18 and 65 years | 32
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: unit was periodontal pocket - one side of the jaw (left or right), not whole patient
  Participants
    Female | 18
    Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants] — Population: unit was periodontal pocket - one side of the jaw (left or right), not whole patient
  participants
    Serbia | 32
mean value of periodontal pockets on one side of the jaw [Mean (Standard Deviation); unit: periodontal pocket] | 32 (0)

OUTCOME MEASURES:

1. Primary Outcome: Periodontal Pocket Depth-PPD
Description: assessment of periodontal pocket depth by probing, mean value of periodontal pockets on one side of the jaw
Time Frame: baseline measure (before the intervention)
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: periodontal pocket
Groups:
- SRP + Injectable Platelet-Rich Fibrin: The side of the mouth which will be treated with scaling and root planing in conjunction with Injectable Platelet-Rich Fibrin
- SRP + Placebo: The side of the mouth which will be treated with scaling and root planing in conjunction with saline
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (periodontal pocket) | 30 | 30
mm | 3.735 (0.863) | 3.696 (0.851)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.429, Wilcoxon (Mann-Whitney) — p<0.05

2. Primary Outcome: Periodontal Pocket Depth-PPD - 1m
Description: assessment of periodontal pocket depth by probing, mean value of periodontal pockets on one side of the jaw
Time Frame: after 1 month
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: periodontal pocket
Groups:
- SRP + Injectable Platelet-Rich Fibrin: Scaling and root planing in conjunction with Injectable Platelet-Rich Fibrin
  SRP + Injectable Platelet-Rich Fibrin: Injectable Platelet-Rich Fibrin application as adjunct to scaling and root planing at baseline - the assessment after 1 month.
- SRP + Placebo: Scaling and root planing in conjunction with saline
  SRP + placebo: Saline application during scaling and root planing at baseline. The assessment after 1 month.
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (periodontal pocket) | 30 | 30
mm | 2.398 (0.792) | 2.876 (0.804)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney) — p<0.05

3. Primary Outcome: Periodontal Pocket Depth-PPD - 3m
Description: assessment of periodontal pocket depth by probing, mean value of periodontal pockets on one side of the jaw
Time Frame: after 3 months
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: periodontal pocket
Groups:
- SRP + Injectable Platelet-Rich Fibrin: Scaling and root planing in conjunction with Injectable Platelet-Rich Fibrin
  SRP + Injectable Platelet-Rich Fibrin: Injectable Platelet-Rich Fibrin application as adjunct to scaling and root planing at baseline - the assessment after 3 months.
- SRP + Placebo: Scaling and root planing in conjunction with saline
  SRP + placebo: Saline application during scaling and root planing at baseline - the assessment after 3 months.
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (periodontal pocket) | 30 | 30
mm | 1.990 (0.640) | 2.567 (0.701)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney) — p<0.05

4. Primary Outcome: Periodontal Pocket Depth-PPD - 6
Description: assessment of periodontal pocket depth by probing mean value of one side of the jaw
Time Frame: after 6 months
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: periodontal pocket
Groups:
- SRP + Injectable Platelet-Rich Fibrin: Scaling and root planing in conjunction with Injectable Platelet-Rich Fibrin
  SRP + Injectable Platelet-Rich Fibrin: Injectable Platelet-Rich Fibrin application as adjunct to scaling and root planing at baseline - the assessment after 6 month.
- SRP + Placebo: Scaling and root planing in conjunction with saline
  SRP + placebo: Saline application during scaling and root planing at baseline. The assessment after 6 month.
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (periodontal pocket) | 30 | 30
mm | 1.778 (0.542) | 2.409 (0.640)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney) — p<0.05

5. Primary Outcome: Level of Gingival Margin-LGM
Description: assessment of level of gingival margin-LGM by probing, i.e.distance between cementoenamel junction and gingival margin (the most coronal point of the gingiva); mean value of one side of the jaw
Time Frame: baseline measure (before the intervention)
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: periodontal pocket
Groups:
- SRP + Injectable Platelet-Rich Fibrin: The side of the mouth which will be treated with scaling and root planing in conjunction with Injectable Platelet-Rich Fibrin SRP + Injectable Platelet-Rich Fibrin: Injectable Platelet-Rich Fibrin application as adjunct to scaling and root planing
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (periodontal pocket) | 30 | 30
mm | 1.737 (0.567) | 1.787 (0.589)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.575, Wilcoxon (Mann-Whitney) — p<0.05

6. Primary Outcome: Level of Gingival Margin-LGM - 1m
Description: as for outcome 5
Time Frame: after 1 month
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: periodontal pocket
Groups:
- SRP + Placebo: Scaling and root planing in conjunction with saline
  SRP + placebo: Saline application during scaling and root planing at baseline - the assessment after 1 month.
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (periodontal pocket) | 30 | 30
mm | 0.948 (0.573) | 1.150 (0.462)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.575, Wilcoxon (Mann-Whitney) — p<0.05

7. Primary Outcome: Level of Gingival Margin-LGM - 3m
Description: assessment of level of gingival margin-LGM by probing, i.e. distance between cementoenamel junction and gingival margin (the most coronal point of the gingiva); mean value of one side of the jaw
Time Frame: after 3 months
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: periodontal pocket
Groups:
- SRP + Placebo: Scaling and root planing in conjunction with saline
  SRP + placebo: Saline application during scaling and root planing at baseline -the assessment after 3 months.
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (periodontal pocket) | 30 | 30
mm | 0.782 (0.580) | 0.877 (0.533)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.249, Wilcoxon (Mann-Whitney) — p<0.05

8. Primary Outcome: Level of Gingival Margin-LGM - 6m
Description: assessment of level of gingival margin-LGM by probing, distance between cementoenamel junction and gingival margin (the most coronal point of the gingiva) after 6 months
Time Frame: after 6 months
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: periodontal pocket
Groups:
- SRP + Injectable Platelet-Rich Fibrin: Scaling and root planing in conjunction with Injectable Platelet-Rich Fibrin
  SRP + Injectable Platelet-Rich Fibrin: Injectable Platelet-Rich Fibrin application as adjunct to scaling and root planing at baseline - the assessment after 6 months.
- SRP + Placebo: Scaling and root planing in conjunction with saline
  SRP + placebo: Saline application during scaling and root planing at baseline. The assessment after 6 months.
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (periodontal pocket) | 30 | 30
mm | 0.808 (0.518) | 0.794 (0.457)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.871, Wilcoxon (Mann-Whitney) — p<0.05

9. Primary Outcome: Clinical Attachment Level- CAL
Description: assessment of clinical attachment level- CAL by probing
Time Frame: baseline measure (before the intervention)
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (periodontal pocket) | 30 | 30
mm | 2.009 (0.724) | 2.018 (0.715)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.773, Wilcoxon (Mann-Whitney) — p<0.05

10. Primary Outcome: Clinical Attachment Level- CAL - 1m
Description: assessment of clinical attachment level- CAL by probing, mean value of one side of the jaw
Time Frame: after 1 month
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (periodontal pocket) | 30 | 30
mm | 1.453 (0.643) | 1.755 (0.654)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney) — p<0.05

11. Primary Outcome: Clinical Attachment Level- CAL - 3m
Description: assessment of clinical attachment level- CAL by probing, mean value of one side of the jaw
Time Frame: after 3 months
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (periodontal pocket) | 30 | 30
mm | 1.237 (0.610) | 1.619 (0.618)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney) — p<0.05; p<0.05

12. Primary Outcome: Clinical Attachment Level- CAL - 6m
Description: assessment of clinical attachment level- CAL by probing, mean value of one side of the jaw
Time Frame: after 6 months
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (periodontal pocket) | 30 | 30
mm | 1.226 (0.580) | 1.585 (0.619)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney) — p<0.05

13. Primary Outcome: Bleeding on Probing-BOP
Description: assessment of bleeding on probing Mühlemann Papillary Bleeding Index , a four-grade index based on both the extent of bleeding and the time it takes for bleeding to occur after stimulation with a periodontal probe (0-the best outcome, 4-the worst outcome).
Time Frame: baseline measure (before the intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (periodontal pocket) | 30 | 30
score on a scale | 1.418 (0.714) | 1.345 (0.711)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.063, Wilcoxon (Mann-Whitney) — p<0.05

14. Primary Outcome: Bleeding on Probing-BOP - 1m
Description: as for outcome 13
Time Frame: after 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (periodontal pocket) | 30 | 30
score on a scale | 0.649 (0.454) | 1.005 (0.562)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney) — p<0.05

15. Primary Outcome: Bleeding on Probing-BOP 3m
Description: as for outcome 13
Time Frame: after 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (periodontal pocket) | 30 | 30
score on a scale | 0.298 (0.280) | 0.601 (0.392)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney) — p<0.05

16. Primary Outcome: Bleeding on Probing-BOP - 6m
Description: as for outcome 13
Time Frame: after 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (periodontal pocket) | 30 | 30
score on a scale | 0.098 (0.090) | 0.257 (0.167)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney) — p<0.05

17. Primary Outcome: Plaque Index- PI
Description: visual assessment of plaque index-PI and by probing Plaque Index (Silness and Löe), 0-the best outcome, 3-the worst outcome
Time Frame: baseline measure (before the intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (periodontal pocket) | 30 | 30
score on a scale | 1.231 (0.559) | 1.241 (0.565)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.085, Wilcoxon (Mann-Whitney) — p<0.05

18. Primary Outcome: Plaque Index- PI -1m
Description: as for outcome 17
Time Frame: after 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (periodontal pocket) | 30 | 30
score on a scale | 0.255 (0.202) | 0.250 (0.185)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney) — p<0.05

19. Primary Outcome: Plaque Index- PI -3m
Description: as for outcome 17
Time Frame: after 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (periodontal pocket) | 30 | 30
score on a scale | 0.236 (0.254) | 0.212 (0.182)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney) — p<0.05

20. Primary Outcome: Plaque Index- PI - 6m
Description: visual assessment of plaque index-PI and by probing
Time Frame: after 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (periodontal pocket) | 30 | 30
score on a scale | 0.199 (0.185) | 0.203 (0.184)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.895, Wilcoxon (Mann-Whitney) — p<0.05

21. Primary Outcome: Number of Periodontal Pockets With Presence/Absence of Aggregatibacter Actinomycetemcomitans (Aa) in Gingival Crevicular Fluid (GCF)
Description: Number of periodontal pockets with presence/absence of Aggregatibacter actinomycetemcomitans in gingival crevicular fluid (GCF) at baseline
Time Frame: baseline measure (before the intervention)
Measure: Count of Units; unit: GCF- periodontal pocket
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
GCF- periodontal pocket
  Presence of microorganism | 24 | 24
  Absence of mimcroorganism | 6 | 6
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.999, McNemar — p<0.05

22. Primary Outcome: Number of Periodontal Pockets With Presence/Absence of Aggregatibacter Actinomycetemcomitans (Aa) in Gingival Crevicular Fluid (GCF) -1m
Description: Number of periodontal pockets with presence/absence of Aggregatibacter actinomycetemcomitans in gingival crevicular fluid (GCF) after 1 month
Time Frame: after 1 month
Measure: Count of Units; unit: GCF- periodontal pocket
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
GCF- periodontal pocket
  Presence of microorganism | 5 | 18
  Absence of mimcroorganism | 25 | 12
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, McNemar — p<0.05

23. Primary Outcome: Number of Periodontal Pockets With Presence/Absence of Aggregatibacter Actinomycetemcomitans (Aa) in Gingival Crevicular Fluid (GCF) - 3m
Description: Number of periodontal pockets with presence/absence of Aggregatibacter Actinomycetemcomitans (Aa) in Gingival Crevicular Fluid (GCF) after 3 months
Time Frame: after 3 months
Measure: Count of Units; unit: GCF- periodontal pocket
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
GCF- periodontal pocket
  Presence of microorganism | 8 | 16
  Absence of mimcroorganism | 22 | 14
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.008, McNemar — p<0.05

24. Primary Outcome: Number of Periodontal Pockets With Presence/Absence of Aggregatibacter Actinomycetemcomitans (Aa) in Gingival Crevicular Fluid (GCF) - 6m
Description: Number of periodontal pockets with presence/absence of Aggregatibacter actinomycetemcomitans in gingival crevicular fluid (GCF) after 6 months
Time Frame: after 6 months
Measure: Count of Units; unit: GCF- periodontal pocket
Units Other Than Participants: GCF- periodontal pocket
Groups:
- SRP + Placebo: Scaling and root planing in conjunction with saline
  SRP + placebo: Saline application during scaling and root planing at baseline - the assessment after 6 months
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
GCF- periodontal pocket
  Presence of microorganism | 17 | 19
  Absence of mimcroorganism | 13 | 11
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.500, McNemar — p<0.05

25. Primary Outcome: Number of Periodontal Pockets With Presence/Absence of Porphyromonas Gingivalis (Pg) in Gingival Crevicular Fluid (GCF)
Description: Number of periodontal pockets with presence/absence of Porphyromonas gingivalis - Pg in gingival crevicular fluid (GCF) at baseline
Time Frame: baseline measure (before the intervention)
Measure: Count of Units; unit: GCF- periodontal pocket
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
GCF- periodontal pocket
  Presence of microorganism | 30 | 30
  Absence of mimcroorganism | 0 | 0
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.999, McNemar — p<0.05

26. Primary Outcome: Number of Periodontal Pockets With Presence/Absence of Porphyromonas Gingivalis (Pg) in Gingival Crevicular Fluid (GCF) - 1m
Description: Number of periodontal pockets with presence/absence of Porphyromonas gingivalis - Pg in gingival crevicular fluid (GCF) after 1 month
Time Frame: after 1 month
Measure: Count of Units; unit: GCF- periodontal pocket
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
GCF- periodontal pocket
  Presence of microorganism | 12 | 28
  Absence of mimcroorganism | 18 | 2
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, McNemar — p<0.05

27. Primary Outcome: Number of Periodontal Pockets With Presence/Absence of Porphyromonas Gingivalis (Pg) in Gingival Crevicular Fluid (GCF) - 3m
Description: Number of periodontal pockets with presence/absence of Porphyromonas gingivalis - Pg in gingival crevicular fluid after 3 months.
Time Frame: after 3 months
Measure: Count of Units; unit: GCF- periodontal pocket
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
GCF- periodontal pocket
  Presence of microorganism | 21 | 27
  Absence of mimcroorganism | 9 | 3
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.40, McNemar — p<0.05

28. Primary Outcome: Number of Periodontal Pockets With Presence/Absence of Porphyromonas Gingivalis (Pg) in Gingival Crevicular Fluid (GCF) - 6m
Description: Number of periodontal pockets with presence/absence of Porphyromonas gingivalis - Pg in gingival crevicular fluid after 6 months.
Time Frame: after 6 months
Measure: Count of Units; unit: GCF- periodontal pocket
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
GCF- periodontal pocket
  Presence of microorganism | 28 | 29
  Absence of mimcroorganism | 2 | 1
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.999, McNemar

29. Primary Outcome: Number of Periodontal Pockets With Presence/Absence of Prevotella Intermedia (Pi) in Gingival Crevicular Fluid (GCF)
Description: Number of periodontal pockets with presence/absence of Prevotella intermedia-Pi in gingival crevicular fluid (GCF) at baseline
Time Frame: baseline measure (before the intervention)
Measure: Count of Units; unit: GCF- periodontal pocket
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
GCF- periodontal pocket
  Presence of microorganism | 27 | 27
  Absence of mimcroorganism | 3 | 3
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.999, McNemar — p<0.05

30. Primary Outcome: Number of Periodontal Pockets With Presence/Absence of Prevotella Intermedia (Pi) in Gingival Crevicular Fluid (GCF) -1m
Description: Number of periodontal pockets with presence/absence of Prevotella intermedia-Pi in gingival crevicular fluid (GCF) after 1 month.
Time Frame: after 1 month
Measure: Count of Units; unit: GCF- periodontal pocket
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
GCF- periodontal pocket
  Presence of microorganism | 12 | 23
  Absence of mimcroorganism | 18 | 7
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.001, McNemar — p<0.05

31. Primary Outcome: Number of Periodontal Pockets With Presence/Absence of Prevotella Intermedia (Pi) in Gingival Crevicular Fluid (GCF) - 3m
Description: Number of periodontal pockets with presence/absence of Prevotella intermedia-Pi in gingival crevicular fluid (GCF) after 3 months.
Time Frame: after 3 months
Measure: Count of Units; unit: GCF- periodontal pocket
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
GCF- periodontal pocket
  Presence of microorganism | 17 | 20
  Absence of mimcroorganism | 13 | 10
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.453, McNemar — p<0.05

32. Primary Outcome: Number of Periodontal Pockets With Presence/Absence of Prevotella Intermedia (Pi) in Gingival Crevicular Fluid (GCF) -6m
Description: Number of periodontal pockets with presence/absence of Prevotella intermedia-Pi in gingival crevicular fluid (GCF) after 6 months.
Time Frame: after 6 months
Measure: Count of Units; unit: GCF- periodontal pocket
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
GCF- periodontal pocket
  Presence of microorganism | 22 | 24
  Absence of mimcroorganism | 8 | 6
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.625, McNemar — p<0.05

33. Primary Outcome: Number of Periodontal Pockets With Presence/Absence of Tannerella Forsythia (Tf) in Gingival Crevicular Fluid (GCF)
Description: Number of periodontal pockets with presence/absence of Tannerella forsythia-Tf in gingival crevicular fluid (GCF) at baseline
Time Frame: baseline measure (before the intervention)
Measure: Count of Units; unit: GCF- periodontal pocket
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
GCF- periodontal pocket
  Presence of microorganism | 24 | 24
  Absence of mimcroorganism | 6 | 6
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.999, McNemar

34. Primary Outcome: Number of Periodontal Pockets With Presence/Absence of Tannerella Forsythia (Tf) in Gingival Crevicular Fluid (GCF) - 1m
Description: Number of periodontal pockets with presence/absence of Tannerella forsythia-Tf in gingival crevicular fluid (GCF) after 1 month.
Time Frame: after 1 month
Measure: Count of Units; unit: GCF- periodontal pocket
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
GCF- periodontal pocket
  Presence of microorganism | 7 | 23
  Absence of mimcroorganism | 23 | 7
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, McNemar — p<0.05

35. Primary Outcome: Number of Periodontal Pockets With Presence/Absence of Tannerella Forsythia (Tf) in Gingival Crevicular Fluid (GCF) - 3m
Description: Number of periodontal pockets with presence/absence of Tannerella forsythia-Tf in gingival crevicular fluid (GCF) after 3 months.
Time Frame: after 3 months
Measure: Count of Units; unit: GCF- periodontal pocket
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
GCF- periodontal pocket
  Presence of microorganism | 11 | 24
  Absence of mimcroorganism | 19 | 6
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.001, McNemar — p<0.05

36. Primary Outcome: Number of Periodontal Pockets With Presence/Absence of Tannerella Forsythia (Tf) in Gingival Crevicular Fluid (GCF) - 6m
Description: Number of periodontal pockets with presence/absence of Tannerella forsythia-Tf in gingival crevicular fluid (GCF) after 6 months.
Time Frame: after 6 months
Measure: Count of Units; unit: GCF- periodontal pocket
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
GCF- periodontal pocket
  Presence of microorganism | 17 | 24
  Absence of mimcroorganism | 13 | 6
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.065, McNemar — p<0.05

37. Primary Outcome: Periodontal Pocket Microorganisms
Description: The concentration of periodontal pocket microorganisms determined in gingival crevicular fluid (GCF) by qPCR-real time.
Time Frame: baseline measure (before the intervention)
Measure: Mean (Standard Deviation); unit: copy number
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
copy number | 2408369.00 (3488796.726) | 2372881.00 (3483340.472)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.821, Wilcoxon (Mann-Whitney) — p<0.05

38. Primary Outcome: Periodontal Pocket Microorganisms -1m
Description: The concentration of periodontal pocket microorganisms determined in gingival crevicular fluid (GCF) by qPCR-real time after 1 month.
Time Frame: after 1 month
Measure: Mean (Standard Deviation); unit: copy number
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
copy number | 27708.86 (60036.838) | 323142 (458640)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney) — p<0.05

39. Primary Outcome: Periodontal Pocket Microorganisms - 3m
Description: The concentration of periodontal pocket microorganisms determined in gingival crevicular fluid (GCF) by qPCR-real time after 3 months.
Time Frame: after 3 months
Measure: Mean (Standard Deviation); unit: copy number
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
copy number | 825098.93 (4246296.647) | 226048.10 (680604)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney) — p<0.05

40. Primary Outcome: Periodontal Pocket Microorganisms - 6m
Description: The concentration of periodontal pocket microorganisms determined in gingival crevicular fluid (GCF) by qPCR-real time after 6 months.
Time Frame: after 6 months
Measure: Mean (Standard Deviation); unit: copy number
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
copy number | 71493.73 (95627.954) | 336812.27 (1057691)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney) — p<0.05

41. Primary Outcome: Tumor Necrosis Factor Alpha-TNF-α
Description: concentration of Tumor necrosis factor alpha-TNF-α in GCF using ELISA Kit
Time Frame: baseline measure (before the intervention)
Measure: Mean (Standard Deviation); unit: pg/µl
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
pg/µl | 0.925 (0.109) | 0.918 (0.105)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney) — p<0.05

42. Primary Outcome: Tumor Necrosis Factor Alpha-TNF-α -1m
Description: The concentration of Tumor necrosis factor alpha-TNF-α in GCF using ELISA Kit
Time Frame: after 1 month
Measure: Mean (Standard Deviation); unit: pg/µl
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
pg/µl | 0.382 (0.040) | 0.782 (0.092)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney) — p<0.05

43. Primary Outcome: Tumor Necrosis Factor Alpha-TNF-α - 3m
Description: The concentration of Tumor necrosis factor alpha-TNF-α using ELISA Kit after 3 months.
Time Frame: after 3 months
Measure: Mean (Standard Deviation); unit: pg/µl
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
pg/µl | 0.259 (0.040) | 0.587 (0.104)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney) — p<0.05

44. Primary Outcome: Tumor Necrosis Factor Alpha-TNF-α -6m
Description: The concentration of Tumor necrosis factor alpha-TNF-α using ELISA Kit after 6 months.
Time Frame: after 6 months
Measure: Mean (Standard Deviation); unit: pg/µl
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
pg/µl | 0.238 (0.034) | 0.456 (0.072)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney)

45. Primary Outcome: Matrix Metalloproteinase 8 - MMP-8
Description: The concentration of Matrix metalloproteinase 8 - MMP-8 in GCF using ELISA Kit
Time Frame: baseline measure (before the intervention)
Measure: Mean (Standard Deviation); unit: pg/ml
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
pg/ml | 11.315 (1.741) | 11.336 (1.720)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.671, Wilcoxon (Mann-Whitney) — p<0.05

46. Primary Outcome: Matrix Metalloproteinase 8 - MMP-8 -1m
Description: The concentration of Matrix metalloproteinase 8 - MMP-8 in GCF using ELISA Kit after 1 month.
Time Frame: after 1 month
Measure: Mean (Standard Deviation); unit: pg/ml
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
pg/ml | 7.906 (1.356) | 9.964 (1.488)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney) — p<0.05

47. Primary Outcome: Matrix Metalloproteinase 8 - MMP-8 - 3m
Description: The concentration of Matrix metalloproteinase 8 - MMP-8 using ELISA Kit after 3 months.
Time Frame: after 3 months
Measure: Mean (Standard Deviation); unit: pg/ml
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
pg/ml | 6.010 (1.357) | 9.061 (1.364)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney) — p<0.05

48. Primary Outcome: Matrix Metalloproteinase 8 - MMP-8 - 6m
Description: The concentration of Matrix metalloproteinase 8 - MMP-8 using ELISA Kit after 6 months.
Time Frame: after 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
pg/ml | 4.681 (1.465) | 8.642 (1.303)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney)

49. Primary Outcome: Alkaline Phosphatase - ALP
Description: The concentration of Alkaline phosphatase - ALP in GCF using ELISA Kit
Time Frame: baseline measure (before the intervention)
Measure: Mean (Standard Deviation); unit: pg/ml
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
pg/ml | 280.496 (95.941) | 280.852 (96.263)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.753, Wilcoxon (Mann-Whitney) — p<0.05

50. Primary Outcome: Alkaline Phosphatase - ALP -1m
Description: The concentration of Alkaline phosphatase - ALP in GCF using ELISA Kit after 1 month.
Time Frame: after 1 month
Measure: Mean (Standard Deviation); unit: pg/ml
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
pg/ml | 116.936 (37.529) | 199.666 (76.413)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney) — p<0.05

51. Primary Outcome: Alkaline Phosphatase - ALP -3m
Description: The concentration of Alkaline phosphatase - ALP using ELISA Kitafter 3 months.
Time Frame: after 3 months
Measure: Mean (Standard Deviation); unit: pg/ml
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
pg/ml | 145.716 (49.959) | 216.835 (79.486)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney) — p<0.05

52. Primary Outcome: Alkaline Phosphatase - ALP -6m
Description: The concentration of Alkaline phosphatase - ALP using ELISA Kit after 6 months.
Time Frame: after 6 months
Measure: Mean (Standard Deviation); unit: pg/ml
Units Other Than Participants: GCF- periodontal pocket
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
Number analyzed (Participants) | 30 | 30
Number analyzed (GCF- periodontal pocket) | 30 | 30
pg/ml | 237.554 (79.872) | 268.905 (90.331)
Statistical Analysis 1: Comparison: SRP + Injectable Platelet-Rich Fibrin vs SRP + Placebo; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney) — p<0.05

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored/assessed.
Description: Adverse events were not monitored/assessed.
Groups:
- SRP + Placebo: Scaling and root planing in conjunction with saline
  SRP + placebo: Saline as adjunct to scaling and root planing
Arm/Group | SRP + Injectable Platelet-Rich Fibrin | SRP + Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-04-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT04178590/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT04178590/SAP_001.pdf
  • Informed Consent Form (2020-04-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT04178590/ICF_002.pdf